CLINICAL TRIAL: NCT02661035
Title: Allogeneic Hematopoietic Stem Cell Transplantation Using Reduced Intensity Conditioning (RIC) for the Treatment of Hematological Diseases [MT2015-32]
Brief Title: Allo HSCT Using RIC for Hematological Diseases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015LS152
Record Dates: First submitted 2016-01-19; First posted 2016-01-21 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Acute Myelogenous Leukemia; Acute Lymphocytic Leukemia; Chronic Myelogenous Leukemia; Plasma Cell Leukemia; Myelodysplastic Syndromes; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; B-Cell Lymphoma; Follicular Lymphoma; Lymphoplasmacytic Lymphoma; Mantle-Cell Lymphoma; Prolymphocytic Leukemia; Lymphoblastic Lymphoma; Burkitt's Lymphoma; Non-Hodgkin's Lymphoma; Multiple Myeloma; Myeloproliferative Syndromes; Hematological Diseases
Keywords: AML; ALL; CML; MDS; CLL; SLL; NHL
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Plasma Cell; Myelodysplastic Syndromes; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell; Leukemia, Prolymphocytic; Burkitt Lymphoma; Lymphoma, Non-Hodgkin; Multiple Myeloma; Hematologic Diseases | interventions — Allopurinol; fludarabine; fludarabine phosphate; Cyclophosphamide; Antilymphocyte Serum; Whole-Body Irradiation; Tacrolimus; Mycophenolic Acid; Association

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reduced Intensity Conditioning (Experimental): Non-myeloablative cyclophosphamide/ fludarabine/total body irradiation (TBI) preparative regimen followed by a related or unrelated donor stem cell infusion
  Interventions: Drug: Allopurinol; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: ATG; Radiation: TBI; Drug: Tacrolimus; Drug: MMF; Biological: Peripheral Blood Stem Cells; Biological: Related or Unrelated Bone Marrow Cells

INTERVENTIONS:
Drug: Allopurinol — 300 mg/day (for peds -150 mg/m^2/day), day -6 and continue through day 0 or longer if clinically indicated
  Other Names: Zyloprim
Drug: Fludarabine — 30 mg/m^2 IV over 1 hour, day -6, -5, -4, -3 and -2
  Other Names: Fludara
Drug: Cyclophosphamide — 50 mg/kg IV over 2 hours, day -6
  Other Names: Cytoxan
Drug: ATG — Only for patients with an unrelated donor (URD) and NO multi-agent chemotherapy 3 months prior to transplant. ATG will be administered IV every 12 hours for 6 doses on days -6, -5, and -4 according to institutional guidelines. Methylprednisolone 1 mg/kg IV administered immediately prior to each dose of ATG (6 doses).
  Other Names: Anti-thymocyte globulin
Radiation: TBI — All patients who have had previous radiation therapy or TBI will be seen by Radiation Oncology prior to entrance on the protocol for approval for additional 200 cGy of TBI. TBI may be delivered by local guidelines provided the effective dose is equivalent to what is recommended in the TBI Guidelines. The dose of TBI will be 200 cGy given in a single fraction on day -1.
  Other Names: Total body irradiation
Drug: Tacrolimus — All patients will receive tacrolimus therapy beginning on day -3. Initial dosing of tacrolimus will be 0.03 - 0.05 mg/kg/day IV; if the recipient body weight is <40 kg, dosing will be 3 times daily, and if ≥ 40 kg, twice daily or per current institutional guidelines.
  An attempt will be made to maintain a trough level of 5-10 ng/mL and subsequent dose modifications will be provided by the pharmacist.
  Once the patient can tolerate oral medications and has a reasonable oral intake, tacrolimus will be converted to an oral form based on the current IV dose providing normal renal and hepatic function and no major drug interactions.
  The timing of the tacrolimus taper will be at the discretion of the treating physician, but in general:
  * Taper begins at day +100 +/- 10 days, if the patient is stably engrafted and has no active GVHD.
  * Taper to zero by reducing dose by approximately 10% a week (rounded to nearest pill size), with a goal to discontinue by month 6 post-HCT.
  Other Names: Prograf
Drug: MMF — 3 gram/day IV/PO for patients who are ≥ 40 kg divided in 2 or 3 doses. In obese patients (>125% IBW) 15 mg/kg every 12 hours may be considered. Pediatric patient (<40 kilograms) will receive MMF at the dose of 15 mg/kg/dose every 8 hours beginning day -3. MMF dosing will be monitored and altered as clinically appropriate based on institutional guidelines. Patients will be eligible for MMF dosing and pharmacokinetics studies.
  MMF will stop at day +30 or 7 days after engraftment, whichever day is later, if no acute GVHD. (Definition of engraftment is 1st day of 3 consecutive days of absolute neutrophil count [ANC) ≥ 0.5 x 109 /L]). If no donor engraftment, MMF will continue as long as clinically indicated.
  Other Names: Mycophenolate Mofetil
Biological: Peripheral Blood Stem Cells — On day 0, patients will receive an allogeneic transplant using PBSC which are CD34+ selected as the donor graft. The graft will be infused over 15-60 minutes after premedication with acetaminophen 650 mg PO and diphenhydramine 25 mg PO/IV with doses adjusted for pediatric patients.
Biological: Related or Unrelated Bone Marrow Cells — On day 0, a target dose of 3 x 10^8 nucleated cells/kg recipient weight will be collected. The graft will be infused over 15-60 minutes after premedication with acetaminophen 650 mg PO and diphenhydramine 25 mg PO/IV with doses adjusted for pediatric patients.

SUMMARY:
This is a phase II trial using a non-myeloablative cyclophosphamide/ fludarabine/total body irradiation (TBI) preparative regimen followed by a related or unrelated donor stem cell infusion. The primary objective is to evaluate rates of acute graft-versus-host disease (GVHD) grades II-IV and chronic GVHD with an updated GVHD prophylaxis of tacrolimus and mycophenolate mofetil (MMF) with a non-myeloablative preparative regimen in persons with hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Age, Performance Status, and Graft Criteria

  * Age 0 to 70 years of age with Karnofsky score ≥ 70% (≥ 16 years) or Lansky score ≥ 50 (< 16 years)
  * Patients ≥ 70 and ≤ 75 years of age may be eligible if they have a HCT-CI Co-Morbidity score ≤ 2
  * Must be ≥ 3 months after prior myeloablative transplant, if applicable
  * 5/6 or 6/6 related donor match or a 7-8/8 HLA-A,B,C,DRB1 allele matched unrelated donor marrow and/or PBSC donor match per current institutional guidelines Related donors will be evaluated and collected per MT2012-14C; Unrelated donors will be identified and collected per usual procedures
* Eligible Diseases

  * Acute Myeloid Leukemia (AML): high risk CR1 (as evidenced by preceding MDS, high risk cytogenetics, ≥ 2 cycles to obtain CR, erythroblastic or megakaryocytic leukemia, FLT-3 ITD +; CR2+. All patients must be in CR as defined by hematological recovery, AND <5% blasts by light microscopy within the bone marrow with a cellularity of ≥15%.
  * Very high risk pediatric patients with AML: Patients <21 years, however, are eligible with (M2 marrow) with < 25% blasts in marrow after having failed one or more cycles of chemotherapy.
  * Acute Lymphocytic Leukemia (ALL): factor that define high risk CR1 include but are not limited to cytogenetics demonstrating t(9;22), t (1:19), t(4;11), other MLL rearrangements, hypodiploidy, or IKZF1 abnormalities), DNA index < 0.81, > 1 cycle to obtain CR or presence minimal residual disease (MRD). Patients in CR2+ are eligible. All patients must be in CR as defined by hematological recovery, AND <5% blasts by light microscopy within the bone marrow with a cellularity of ≥15%.
  * Very high risk pediatric patients with ALL: patients <21 years are also considered high risk CR1 if they had M2 or M3 marrow at day 42 from the initiation of induction or M3 marrow at the end of induction. They are eligible once they achieved a complete remission.
  * Chronic Myelogenous Leukemia excluding refractory blast crisis: To be eligible in first chronic phase (CP1) patient must have failed or be intolerant to imatinib mesylate.
  * Plasma Cell Leukemia after initial therapy, who achieved at least a partial remission
  * Myelodysplasia (MDS) requiring transplant as defined as: IPSS INT-2 or High Risk; R-IPSS High or Very High; WHO classification: RAEB-1, RAEB-2; Severe Cytopenias: ANC < 0.8, Anemia or thrombocytopenia requiring transfusion; Poor or very poor risk cytogenetics based on IPSS or R-IPSS definitions; therapy-related MDS. Blasts must be < 5% by bone marrow aspirate morphology.
  * Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL), Marginal Zone B-Cell Lymphoma or Follicular Lymphoma are eligible if there was disease progression/relapse within 12 of achieving a partial or complete remission. Patients who had remissions lasting > 12 months, are eligible after at least two prior therapies. Patients with bulky disease (nodal mass greater than 5 cm) should be considered for de-bulking chemotherapy before transplant.
  * Lymphoplasmacytic Lymphoma, Mantle-Cell Lymphoma, Prolymphocytic Leukemia, NK cell malignancies are eligible after initial therapy in CR1+ or PR1+.
  * Large Cell NHL > CR2/> PR2: Patients in CR2/PR2 with initial short remission (<6 months) are eligible.
  * Lymphoblastic Lymphoma, Burkitt's Lymphoma, and other high-grade NHL after initial therapy if stage III/IV in CR1/PR1 or after progression if stage I/II < 1 year.
  * Multiple Myeloma beyond PR2: Patients with chromosome 13 abnormalities, first response lasting less than 6 months, or β-2 microglobulin > 3 mg/L, may be considered for this protocol after initial therapy.
  * Myeloproliferative Syndromes
* Organ Function Criteria Adequate organ function is defined as:

  * Liver: AST and ALT < 5 x upper limit of normal and bilirubin < 3 x upper limit of normal
  * Renal: Creatinine ≤ 2.0 mg/dl (adults) and estimated glomerular filtration rate (GFR) ≥ 40 mL/min (pediatrics). Adults with a creatinine > 1.2 mg/dl or a history of renal dysfunction must have estimated glomerular filtration rate (GFR) > 40 mL/min.
  * Albumin > 2.5 g/dL
  * Cardiac: Absence of decompensated congestive heart failure, or uncontrolled arrhythmia and left ventricular ejection fraction > 35%.
  * Pulmonary: DLCOcorr ≥ 40% predicted, and absence of O2 requirements. For children that are not able to cooperate with PFTs, a pulse oximetry with or without exercise should be attempted. If neither test can be obtained it should be clearly stated in the physician's note.
* If recent mold infection (e.g. aspergillus) must have minimum of 30 days of therapy and responsive disease and be cleared by Infectious Disease
* Females of child bearing potential and sexually active males must agree to use adequate birth control during study treatment
* Voluntary written consent (adult or parent/guardian with presentation of the minor information sheet, if appropriate)

Exclusion Criteria:

* Pregnant or breast feeding. The agents used in this study include Pregnancy Category D: known to cause harm to a fetus. Females of childbearing potential must have a blood test or urine study within 14 days prior to registration to rule out pregnancy.
* Untreated active infection
* Active CNS disease
* Active HIV infection or known HIV positive serology
* Congenital bone marrow failure syndrome
* Previous irradiation that precludes the safe administration of an additional dose of 200 cGy of TBI
* CML in refractory blast crisis
* Intermediate or high grade NHL, mantle cell NHL, and Hodgkin disease that is progressive on salvage therapy. Stable disease is acceptable to move forward provided it is non-bulky.
* Multiple myeloma progressive on salvage chemotherapy

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-05-29 (Actual)

PRIMARY OUTCOMES:
Evaluate rates of acute graft-versus-host disease (GVHD) II-IV | Day 100 post transplant
  Percent of subjects with grade II-IV acute GVHD

SECONDARY OUTCOMES:
Evaluate rates of chronic GVHD | 1 year post transplant
  Percent of subjects with chronic GVHD
Evaluate neutrophil engraftment without ATG (in siblings) | Day 42 post transplant
  Percent of subjects with neutrophil engraftment without ATG (in siblings)
Evaluate neutrophil engraftment with ATG (in unrelated donors) | Day 42 post transplant
  Percent of subjects with neutrophil engraftment with ATG (in unrelated donors)
Evaluate neutrophil engraftment without ATG (in unrelated donors) | Day 42 post transplant
  Percent of subjects with neutrophil engraftment without ATG (in unrelated donors)
Evaluate relapse without ATG (in siblings) - 1 year | 1 year post transplant
  Percent of subjects who relapsed without ATG (in siblings)
Evaluate relapse without ATG (in siblings) - 2 years | 2 years post transplant
  Percent of subjects who relapsed without ATG (in siblings)
Evaluate relapse with ATG (in unrelated donors) - 1 year | 1 year post transplant
  Percent of subjects who relapsed with ATG (in unrelated donors)
Evaluate relapse with ATG (in unrelated donors) - 2 years | 2 years post transplant
  Percent of subjects who relapsed with ATG (in unrelated donors)
Evaluate relapse without ATG (in unrelated donors) - 1 year | 1 year post transplant
  Percent of subjects who relapsed without ATG (in unrelated donors)
Evaluate relapse without ATG (in unrelated donors) - 2 years | 2 years post transplant
  Percent of subjects who relapsed without ATG (in unrelated donors)
Overall survival | Day 100 post transplant
  Percent of surviving subjects
Overall survival | 1 year post transplant
  Percent of surviving subjects
Overall survival | 3 years post transplant
  Percent of surviving subjects
Transplant related mortality (TRM) | Day 100 post transplant
  Percent of subjects with TRM
Transplant related mortality (TRM) | 1 year post transplant
  Percent of subjects with TRM

CONTACTS AND LOCATIONS:
Overall Officials: Erica Warlick, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States